CLINICAL TRIAL: NCT06666166
Title: Exploratory Clinical Study of SHR-A1811 Combined with Apatinib in the Treatment of Advanced Gastric or Gastroesophageal Junction Adenocarcinoma and Colorectal Cancer
Brief Title: SHR-A1811 Combined with Apatinib in the Treatment of Advanced Gastric or Gastroesophageal Junction Adenocarcinoma and Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yunpeng Liu (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yunpeng Liu, Professor, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC-IIT-SHR-A1811-Apa
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Advanced Gastric Carcinoma; Advanced Gastroesophageal Junction Adenocarcinoma; Advanced Colorectal Cancer
Keywords: apatinib; advanced gastric or gastroesophageal junction adenocarcinoma; advanced colorectal cancer; SHR-A1811

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gastric or gastroesophageal junction adenocarcinoma (Experimental)
  Interventions: Drug: SHR-A1811 & Apartinib
- Advanced colorectal cancer (Experimental)
  Interventions: Drug: SHR-A1811 & Apartinib

INTERVENTIONS:
Drug: SHR-A1811 & Apartinib — SHR-A1811 injection will be administered by intravenous infusion. And apatinib will be administered orally.

SUMMARY:
To evaluate the effectiveness and safety of SHR-A1811 combined with apatinib in the treatment of advanced gastric or gastroesophageal junction adenocarcinoma and colorectal cancer.

DETAILED DESCRIPTION:
This is a prospective, dual arm, exploratory clinical research. To evaluate the effectiveness and safety of SHR-A1811 combined with apatinib in the treatment of advanced gastric or gastroesophageal junction adenocarcinoma and colorectal cancer.

Cohort A will enroll subjects with advanced gastric or gastroesophageal junction adenocarcinoma, while Cohort B will enroll subjects with advanced colorectal cancer.

The primary endpoint is objective remission rate (ORR). Secondary endpoints include disease control rate (DCR), duration of remission (DoR), progression-free survival (PFS), overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Participants voluntarily enrolled in this study and signed an informed consent form, were compliant and co-operated with follow-up visits;
2. Age 18-75 years, including 18 and 75 year, male and female;
3. ECOG (Eastern Cooperative Oncology Group) performance status of 0-1;
4. Has a life expectancy of greater than 3 months;
5. Cohort A: Has histologically confirmed diagnosis of unresectable, locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma;
6. Cohort B: Has histologically confirmed diagnosis of unresectable, locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma;
7. There must be a measurable target lesion that meets the RECIST 1.1 criteria;
8. The function of major organs meets the following criteria(not transfused, not using haematopoietic factors and not corrected with drugs within 14 days):

   1. Absolute neutrophil count (ANC) ≥1.5×10^9/L;
   2. PLT ≥100×10^9/L;
   3. Hb≥9g/dL;
   4. ALB≥3.0g/dL;
   5. total bilirubin ≤1.5 x ULN;
   6. ALT/AST ≤ 2.5 x ULN (When there is liver metastasis, ALT/AST ≤ 5 x ULN);
   7. Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CCr) ≥60mL/min (according to Cockcroft-Gault formula);
   8. prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5×ULN;
   9. Echocardiography （ECHO）/Cardiac radionuclide scan （MUGA showed i.LVEF≥50%);
   10. Urine routine results showed that urine protein <1+; For patients with urine protein ≥2+ at baseline, 24-hour urine collection and 24-hour urine protein quantification <1g should be performed.
9. Females of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the first dose and agree to use a highly effective method of contraception for the duration of the study up to 6 months after the last administration of study drug. Male subjects whose partner is a female of childbearing potential must agree to use a highly effective method of contraception for the duration of the study up to 6 months after the last administration of study drug.

Exclusion Criteria:

1. Patients with meningeal metastases; Or patients with brain metastases that have not been treated with surgery or radiation, but those who have been stable for at least one month after treatment and have stopped using steroid drugs (such as 10mg/day prednisone or other equivalent hormones) for more than 2 weeks except;
2. Uncontrolled pleural effusion or ascites;
3. There are serious concomitant diseases: such as serious cardiovascular and cerebrovascular disease, kidney failure, liver failure, hematopoietic disease, endocrine disease, cachexia, etc;
4. Previously received antibody drug conjugate therapy containing topoisomerase I inhibitors, such as trastuzumab deruxtecan (DS-8201), etc; Subjects underwent surgery (except diagnostic surgery), radiotherapy, chemotherapy, macromolecular targeted therapy or immunotherapy within 4 weeks before the first dose of the study drug；Small molecule targeted drugs (including other oral targeted drugs used in clinical trials) whose last dose is less than 5 half-life period or 4 weeks (whichever is shorter) from the first dose; Subjects received palliative radiotherapy or local treatment less than 2 weeks after completion of treatment and before the first dose;
5. Subjects who have been treated with live vaccine or attenuated vaccine within 1 month prior to the first dose;
6. Subjects requiring systemic therapy with corticosteroids (>10 mg/day of prednisone or equivalent) or other immunosuppressive agents within 14 days prior to first dose, excluding nasal spray or inhaled corticosteroids.
7. The toxicity caused by previous anti-tumor treatments has not recovered to ≤ CTCAE grade 1 (excluding hair loss; according to the researcher's judgment, some tolerable chronic grade II toxicity can be excluded);
8. Uncontrolled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg); Active bleeding (such as local active ulcer lesions and fecal occult blood≥ ++), with a history of gastrointestinal bleeding within 6 months;
9. Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5 × ULN), with a tendency to bleed or undergoing thrombolytic or anticoagulant therapy;
10. Subjects were co-administered a potent CYP3A4 or CYP2D6 inhibitor or inducer within 3 weeks prior to first dosing;
11. Factors affecting oral administration of medications such as inability to swallow, chronic diarrhoea and intestinal obstruction;
12. Any active autoimmune disease or history of autoimmune disease (e.g., autoimmune hepatitis, uveitis, enteritis, pituitary gland inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (may be included after hormone replacement therapy)); and skin disorders (e.g., vitiligo, psoriasis, or alopecia) in which asthma has been in complete remission in childhood and has required no intervention in adulthood or in which systemic therapy is not required.subjects with autoimmune mediated hypothyroidism treated with thyroid replacement hormone at a stable dose and type I diabetes patients treated with insulin at a stable dose can be included;
13. Subjects with immunodeficiency disease, such as HIV infection, congenital or acquired immune dysfunction, organ transplantation；
14. Uncontrolled heart clinical symptoms or diseases, such as (1) New York Heart Association class II or higher heart failure; (2) unstable angina pectoris; (3) Myocardial ischaemia within 1 year; (4) Subjects with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
15. Complicated severe infection within 30 days prior to first dose, including but not limited to infection complications that require hospitalization, bacteremia, severe pneumonia, etc; active infections that have received therapeutic intravenous antibiotics within 2 weeks prior to the first dose. Subjects receiving prophylactic antibiotic treatment (such as preventing urinary tract infections) can be enrolled;
16. Subjects with active hepatitis B (HBsAg positive with HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive with HCV-RNA above the lower limit of detection of the analytical method);
17. Evidence of previously clinically significant lung diseases, including but not limited to interstitial pneumonitis, pneumonitis, pulmonary fibrosis and radiographic pneumonia (Excluding radioactive changes do not require treatment), or suspected subjects with this type of diseases founded during the screening period;
18. Allergy to any investigational drug or its excipients;
19. Concomitant other malignancies ≤5 years prior to enrollment, except adequately treatable carcinoma in situ of the cervix, basal cell or squamous epithelial cell skin cancer, localised prostate cancer, and ductal carcinoma;
20. Serious physical or mental illnesses or laboratory abnormalities. Any condition which, in the opinion of the Investigator, may be detrimental to the subject or result in the subject's inability to meet or perform the requirements of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | baseline up to approximately 6 month
  To evaluate the efficacy of anti-tumor

SECONDARY OUTCOMES:
Duration of Response (DOR) | baseline up to approximately 12 months
  To evaluate the efficacy of anti-tumor
Disease control rate (DCR) | baseline up to approximately 6 month
  To evaluate the efficacy of anti-tumor
Progression-free survival (PFS) | baseline up to approximately 6 month
  To evaluate the efficacy of anti-tumor
Overall survival (OS) | baseline up to approximately 12 month
  To evaluate the efficacy of anti-tumor
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From the initiation of the first dose to 28 days after the last dose
  To identify the incidence of AE and SAE in clinical trial

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of China Medical University, Shenyang, China